CLINICAL TRIAL: NCT05680103
Title: Correlation Between Occlussion Types , in Patients With Temporomandibular Disorders. : A Cross Sectional Study
Brief Title: Correlation Between Occlussion Types , in Patients With Temporomandibular Disorders.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Armia Zaki, Principal Investigator, Cairo University
Other Study IDs: occlussion and TMDs
Record Dates: First submitted 2022-12-25; First posted 2023-01-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: lateral cephalometry — lateral x-ray beam to capture lateral cephalometry of patients

SUMMARY:
study to find if there is correlation between occlusion types and TMD or not

DETAILED DESCRIPTION:
The relationship among occlusion, condylar position and temporomandibular disorders (TMDs) has been part of an extensive discussion in the dental field. There is a strong belief that the discrepancy between the centric relation (CR) and the intercuspal position (ICP) could predispose to the presence of TMDs . It was suggested in the past in the earlier studies that TMD is more common among the individuals who have Angle class II and class III , malocclusion , open bite , and cross bite . In the 1990s, studies suggested that some occlusal and skeletal characteristics as anterior open bite, unilateral posterior crossbite, overjet greater than 6-7mm, absence of five or more posterior teeth and CR to maximum intercuspation (MI) discrepancy greater than 2mm could be considered occlusal risk factors for TMDs . In their study, Oyetola et al. reported that 25% of the evaluated TMD patients had malocclusion Yet, recently with studies and systematic reviews , this idea ( alocclusion is the main cause of TMD) started to lose its support, and many studies showed that sensitivity to nociceptive stimulations and psychological factors are of more importance in the etiology of TMD

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 16 years old and below 50
2. Patients with TMD diagnosed (stage 2 Wilkes classification , anterior disc displacement with reduction, )
3. Provided informed consent.
4. No history of systemic condition affecting TMJ
5. No previous orthodontic ttt

Exclusion Criteria:

1. Ear diseases.
2. History of facial trauma.
3. Neurological or oncological disease.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with TMDs and have teeth for dental occlussion
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ADDwR in patients with class III malocclusion | baseline
  lateral cephalometry will be taken for patients with TMDs and then measurements will be done to calculate SNA and SNB to see Prevalence of ADDwR in patients with class III malocclusion

SECONDARY OUTCOMES:
Prevalence of ADDwR in patients with class I and class II malocclusion | baseline
  lateral cephalometry will be taken for patients with TMDs and then measurements will be done to calculate SNA and SNB to see Prevalence of ADDwR in patients with class I and class II malocclusion

REFERENCES:
- [Background] Maizlin ZV, Nutiu N, Dent PB, Vos PM, Fenton DM, Kirby JM, Vora P, Gillies JH, Clement JJ. Displacement of the temporomandibular joint disk: correlation between clinical findings and MRI characteristics. J Can Dent Assoc. 2010;76:a3. PMID 20633336
- [Background] Cai XY, Jin JM, Yang C. Changes in disc position, disc length, and condylar height in the temporomandibular joint with anterior disc displacement: a longitudinal retrospective magnetic resonance imaging study. J Oral Maxillofac Surg. 2011 Nov;69(11):e340-6. doi: 10.1016/j.joms.2011.02.038. Epub 2011 Jul 1. PMID 21723023